CLINICAL TRIAL: NCT01905553
Title: A Phase 1, Open-label, Randomized, 2-period, Crossover, Exploratory Study to Investigate the Effect of Food on the Bioavailability of a Single Dose of SSP-004184SS in Healthy Adult Subjects
Brief Title: The Effect of Food on the Bioavailability of a Single Dose of SSP-004184SS in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SPD602-113
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Results first posted 2014-12-24 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SSP-004184SS (fed) (Experimental): 21.8 mg/kg (oral capsule form) given once on Day 1 under fed conditions
  Interventions: Drug: SSP-004184SS
- SSP-004184SS (fasted) (Experimental): 21.8 mg/kg (oral capsule form) given once on Day 1 under fasted conditions
  Interventions: Drug: SSP-004184SS

INTERVENTIONS:
Drug: SSP-004184SS — Disodium salt
  Other Names: SPD602

SUMMARY:
To assess the effect of food on the pharmacokinetic profile of SSP-004184 compared to administration under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years inclusive at the time of consent. The date of signing informed consent is defined as the beginning of the Screening Period. This inclusion criterion will only be assessed at the Screening Visit.
* Subject is considered "healthy". Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, and urinalysis.
* Serum ferritin >20ng/mL, hemoglobin >125g/l, and erythrocyte indices within normal range of the clinical laboratory at the Screening Visit and on Day -1: packed cell volume, mean corpuscular volume, and mean corpuscular hemoglobin concentration, or deemed not clinically significant by the investigator.
* Subject is willing to comply with any applicable contraceptive requirements of the protocol and is:
* Male, or
* Female of non-childbearing potential (defined as a female who is post-menopausal [amenorrhea for at least 12 consecutive months] or surgically sterile [hysterectomy, bilateral tubal ligation, bilateral oophorectomy, or bilateral salpingectomy]) and at least 6 weeks post-sterilization
* Non-pregnant, non-lactating female
* At least 90 days post-partum or nulliparous (females only).
* An understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Ability to provide written, personally signed, and dated informed consent to participate in the study, in accordance with International Conference on Harmonisation Good Clinical Practice Guideline E6 (1996) and applicable regulations, before completing any study-related procedures.
* Body mass index between 18.5-30.0kg/m² inclusive. This inclusion criterion will be assessed only at the Screening Visit.
* Ability to swallow the investigational product (multiple capsules at 1 time or consecutively 1 capsule at a time).

Exclusion Criteria:

* A clinically significant history or disorder detected during the medical interview/physical examination such as any cardiovascular, bronchopulmonary, gastrointestinal (eg, inflammatory bowel disease, chronic diarrhea), hepatic, biliary (including gall bladder removal), renal, hematological, endocrine, autoimmune, neurological, or psychiatric disease (including depression) or any other medical condition that is capable of altering the absorption, metabolism, or elimination of drugs; or of constituting a risk factor when taking the investigational product in the judgment of the investigator.
* Confirmed systolic blood pressure >139mmHg or <89mmHg, and diastolic blood pressure >89mmHg or <49mmHg.
* Twelve-lead ECG demonstrating QTc >450msec at screening. If QTc exceeds 450msec, the ECG should be repeated 2 more times and the average of the 3 QTc values should be used to determine the subject's eligibility.
* Subject reports any food allergies, celiac disease, or requirements for specific diet (eg, vegan, vegetarian, low fat).
* Acute illness, as judged by the investigator, within 2 weeks of Day 1 of Treatment Period 1.
* Known or suspected intolerance or hypersensitivity to the investigational products, closely related compounds, or any of the stated ingredients.
* History of thyroid disorder that has not been stabilized on thyroid medication or treatment within 3 months of the Screening Visit.
* History of alcohol or other substance abuse within the last year.
* Routine consumption of more than 3 units of caffeine per day or subjects who experience caffeine withdrawal headaches.
* A positive screen for alcohol or drugs of abuse at the Screening Visit.
* Male subjects who consume more than 3 units of alcohol per day. Female subjects who consume more than 2 units of alcohol per day.
* A positive human immunodeficiency virus antibody screen, hepatitis B surface antigen screen, or hepatitis C virus antibody screen.
* Current use of any other medication (including over-the-counter, herbal, or homeopathic preparations) that could affect (improve or worsen) the study evaluations according to the investigator.
* Use of tobacco in any form (eg, smoking or chewing) or other nicotine-containing products in any form (eg, gum, patch) within 30 days prior to Day 1 of Treatment Period 1.
* Donation of blood or blood products (eg, plasma or platelets) within 60 days prior to Day 1 of Treatment Period 1.
* Use of another investigational product within 30 days prior to Day 1 of Treatment Period 1 or active enrollment in another drug or vaccine clinical study.
* Substantial changes in eating habits within 30 days prior to Day 1 of Treatment Period 1, as assessed by the investigator.
* Prior screen failure, randomization, participation, or enrollment in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-08-27 (Actual); Primary Completion 2013-09-24 (Actual); Study Completion 2013-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Clinical Pharmacology of Miami, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SSP-004184SS Fed First: Subjects received a single dose SSP-004184SS 21.8mg/kg on Day 1 administered 30 minutes after starting a standard high-fat, high-calorie breakfast in Treatment Period 1. During Treatment Period 2, subjects received a single-dose administration of 21.8mg/kg of SSP-004184SS under fasted conditions.
- SSP-004184SS Fasted First: Subjects received a single-dose administration of 21.8mg/kg of SSP-004184SS under fasted conditions on Day 1 in Treatment Period 1. During Treatment Period 2, subjects received a single dose SSP-004184SS 21.8mg/kg on Day 1 administered 30 minutes after starting a standard high-fat, high-calorie breakfast.
Period: Period 1
Arm/Group | SSP-004184SS Fed First | SSP-004184SS Fasted First
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0
Period: Period 2
Arm/Group | SSP-004184SS Fed First | SSP-004184SS Fasted First
Started | 5 | 4
Completed | 4 | 4
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Set consists of all subjects who have taken at least 1 dose of investigational product and have at least 1 post-dose safety assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | SSP-004184SS Fed First | SSP-004184SS Fasted First | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42 (10.89) | 35 (7.62) | 38.9 (9.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to Infinity (AUCinf) of SSP-004184 Under Fasted and Fed Conditions
Description: AUCinf is the area under the plasma concentration versus time curve from time 0 to infinity. AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: Study Periods 1 & 2: Within 30 minutes pre-dose, and Post-dose 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 24, 48, 72 hours.
Population: Pharmacokinetic Set: All subjects in the Safety Set for whom the primary pharmacokinetic data were considered sufficient and interpretable.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SSP-004184SS (Fed) | SSP-004184SS (Fasted)
Number analyzed (Participants) | 9 | 9
ng*hr/mL | 112,236.7 (28,804.8) | 154,676.6 (28,185.7)
Statistical Analysis 1: Comparison: SSP-004184SS (Fed) vs SSP-004184SS (Fasted); Test type: Non-Inferiority or Equivalence — The magnitude effect of food on the pharmacokinetic parameters was evaluated by calculating the point estimate and 90% CIs between Treatment A (test treatment, fed) and Treatment B (reference treatment, fasted); Ratio of Geometric LS Means = 0.718, 90% CI 2-sided [0.670 to 0.770]

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Time of the Last Measureable Concentration (AUClast) of SSP-004184 Under Fed and Fasted Conditions
Description: AUClast is the area under the curve from the time of dosing to the last measurable concentration. AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: Study Periods 1 & 2: Within 30 minutes pre-dose, and Post-dose 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 24, 48, 72 hours.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SSP-004184SS (Fed) | SSP-004184SS (Fasted)
Number analyzed (Participants) | 9 | 9
ng*hr/mL | 112,066.1 (28,822.9) | 154,446 (28,066.5)
Statistical Analysis 1: Comparison: SSP-004184SS (Fed) vs SSP-004184SS (Fasted); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric LS Means = 0.718, 90% CI 2-sided [0.670 to 0.769]

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of SSP-004184 Under Fed and Fasted Conditions
Description: Cmax is a term that refers to the maximum (or peak) concentration that a drug achieves in the body after the drug has been administrated.
Time Frame: Study Periods 1 & 2: Within 30 minutes pre-dose, and Post-dose 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 24, 48, 72 hours.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SSP-004184SS (Fed) | SSP-004184SS (Fasted)
Number analyzed (Participants) | 9 | 9
ng/mL | 32,755.6 (11,797.4) | 70,733.3 (9,782.9)
Statistical Analysis 1: Comparison: SSP-004184SS (Fed) vs SSP-004184SS (Fasted); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric LS Means = 0.449, 90% CI 2-sided [0.380 to 0.530]

ADVERSE EVENTS:
Arm/Group | SSP-004184SS (Fed) | SSP-004184SS (Fasted)
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 5/9 | 4/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SSP-004184SS (Fed) (N=9) | SSP-004184SS (Fasted) (N=9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (2)
Chromaturia (Renal and urinary disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.